CLINICAL TRIAL: NCT07235085
Title: A Phase 3, Multicenter, Double-Masked, Randomized, 3-Arm Parallel Group Study to Evaluate the Efficacy and Safety of Intravitreal OTXTKI (Axitinib Implant) in Participants With Non-Proliferative Diabetic Retinopathy
Brief Title: A Study to Evaluate the Efficacy and Safety of OTX-TKI (Axitinib Implant) in Participants With Non-Proliferative Diabetic Retinopathy
Acronym: HELIOS-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTX-TKI-2025-NPDR-302
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non-Proliferative Diabetic Retinopathy
Keywords: Non-Proliferative Diabetic Retinopathy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OTX-TKI Q52W (single dose) (Experimental): OTX-TKI 0.45 mg via intravitreal (IVT) administration at Day 1 and sham procedure at Week 24
  Interventions: Drug: Single intravitreal injection of axitinib hydrogel implant followed by a mock (sham) injection procedure at Week 24
- OTX-TKI Q24W (2 doses) (Experimental): OTX-TKI 0.45 mg via IVT administration at Day 1 and Week 24
  Interventions: Drug: Intravitreal injection of axitinib hydrogel implant followed by a second intravitreal injection of the axitinib implant at Week 24
- Sham Q24W (control) (Sham Comparator): Sham procedure at Day 1 and Week 24
  Interventions: Other: Sham/mock procedure of intravitreal injection followed by a second sham/mock procedure at Week 24

INTERVENTIONS:
Drug: Single intravitreal injection of axitinib hydrogel implant followed by a mock (sham) injection procedure at Week 24 — OTX-TKI 0.45 mg is a dried polyethylene glycol (PEG)-based hydrogel containing dispersed drug particles of the small molecule axitinib, a tyrosine kinase inhibitor (TKI).
  Arms: OTX-TKI Q52W (single dose)
Drug: Intravitreal injection of axitinib hydrogel implant followed by a second intravitreal injection of the axitinib implant at Week 24 — OTX-TKI 0.45 mg is a dried polyethylene glycol (PEG)-based hydrogel containing dispersed drug particles of the small molecule axitinib, a tyrosine kinase inhibitor (TKI).
  Arms: OTX-TKI Q24W (2 doses)
Other: Sham/mock procedure of intravitreal injection followed by a second sham/mock procedure at Week 24 — sham/mock intravitreal injection procedure
  Arms: Sham Q24W (control)

SUMMARY:
The purpose of this trial is to study the safety and effectiveness of OTX-TKI (axitinib intravitreal hydrogel) for the treatment of Non-Proliferative Diabetic Retinopathy.

OTX-TKI is an intravitreal hydrogel embedded with axitinib. When the OTX-TKI hydrogel is administered into the vitreous cavity of the eye, the hydrogel begins to slowly break down, which allows the axitinib to be slowly released over time.

This clinical trial is comparing OTX-TKI to a "sham" injection procedure. The sham injection is a mock injection procedure, but nothing will actually be inserted in the eye as there is no needle on the sham injector. Only one eye ("study eye") will be treated with study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who is at least 18 years of age at the time of signing the informed consent form (ICF)
2. History of or newly diagnosed with type 1 or 2 diabetes mellitus and have moderately severe to severe NPDR (DRSS levels 47 or 53), confirmed by the Central Reading Center (CRC) based on the images obtained at the Screening visit
3. BCVA Early Treatment Diabetic Retinopathy Study (ETDRS) letter score of ≥ 69 letters (approximate Snellen equivalent of 20/40 or better) in the study eye
4. Willing and able to comply with clinic visits and study-related procedures
5. Provide signed informed consent

Exclusion Criteria:

1. Presence of center-involved diabetic macular edema (CI-DME) defined per protocol via optical coherence tomography (SD-OCT) in the study eye, obtained at the Screening visit
2. Evidence of a rhegmatogenous retinal detachment or visually significant/severe epiretinal membrane, vitreomacular traction syndrome, macular hole, tear of the retinal pigment epithelium in the macula, or other macular pathology in the study eye deemed visually significant by the Investigator
3. In the study eye, any panretinal photocoagulation (PRP) treatment prior to baseline, or received focal or grid laser photocoagulation within 1000 microns of the central subfield of the macula within 6 months prior to baseline
4. IVT anti-VEGF treatment in the study eye within 6 months or port delivery system (PDS) with ranibizumab in the study eye at any time prior to baseline (Day 1)
5. (There are additional exclusion criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
DRSS 2-step change status at Week 52 from baseline in the study eye (≥ 2 step improvement, ≥ 2-step worsening, < 2-step change in either direction) | 52 weeks
  The Diabetic Retinopathy Severity Scale (DRSS) measures the severity of the diabetic retinopathy in patients by grading retinal images obtained by color fundus photography. Severity is determined by the presence of specific signs.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Hu, MD, Principal Investigator — Cumberland Valley Retina Consultants
Locations (1):
- Cumberland Valley Retina Consultants, Hagerstown, Maryland, United States